CLINICAL TRIAL: NCT06504043
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Center Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of HST101 in Healthy Chinese Study Participants With Elevated LDL-C Levels
Brief Title: A Study on Evaluating the Safety of HST101 in Healthy Chinese Participants
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Hasten Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HST101-101
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hypercholesterolemia; Healthy Volunteers; LDL-Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: the initially enrolled 15 subjects will receive low-dose single SC administration, followed by another 15 subjects will receive high-dose single SC administration.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental: cohort low dose HST101 (Experimental): HST101 single SC administration of 150 mg or placebo;
  Interventions: Drug: HST101
- Experimental: cohort high dose HST101 (Experimental): HST101 single SC administration of 300 mg or placebo.
  Interventions: Drug: HST101

INTERVENTIONS:
Drug: HST101 — HST101 is a novel anti-PCSK9 fusion protein
  Other Names: Lerodalcibep

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single HST101 SC dose cohort study to evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Chinese Participants with Elevated LDL-C Levels.

DETAILED DESCRIPTION:
The planned 30 study participants will be assigned to low- or high-dose 2 cohorts and 15 participants in each cohort will be randomized to either the HST101 group or the matching dose placebo group and will be administered in subsequent or in-parallel manner. Cohort 1: 15 study participants will receive the low dose of HST101 or placebo at a corresponding dose. Cohort 2: additional 15 study participants will receive the high dose of HST101 or placebo at a corresponding dose.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are ≥18 and ≤55 years of age with elevated LDL-C Levels;
* LDL-C ≥ 2.6 mmol/L (100 mg/dL) and ≤ 4.9 mmol/L (190 mg/dL) and TG ≤ 2.83 mmol/L (250 mg/dL) who are not on a lipid-lowering therapy 30 days prior to screening;
* Body mass index (BMI) ≥18 and≤28 kg/m2

Exclusion Criteria:

* Positive blood screen for HIV antibody, Treponema pallidum antibody, HBsAg or HCV antibody;
* Clinically significant liver function test abnormalities at screening, such as AST or ALT > 2 × ULN, total bilirubin > 1.5 × ULN, or ALP > 2 × ULN based on normal values;
* CK > 3 × ULN at the screening visit, it can be retested if considered to be related to exercise;
* History of prescription drug abuse, illicit drug use or alcohol abuse;
* Use of any prescription drug, herbal and compound decoction, vitamins, minerals, and OTC drugs and nutritional supplements that alter lipid metabolism within 14 days prior to Check-in and planned use of the above drugs throughout the study;
* Prior treatment with PCSK9 inhibitors, including mAbs, siRNA products, or any Adnectin products;
* History of allergy to protein-based biologics including, but not limited to, mAbs and vaccine;
* Less than 30 days or less than 5 half-lives (drug) since the end of participation in another clinical trial (drug or device), whichever is longer;
* Use of any other biologics within 3 months prior to investigational product administration;
* Any other significant clinical diseases or psychological diseases that the investigator considers to be inappropriate for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety and tolerability of a single SC dose of HST101 in Chinese healthy adult study participants with elevated LDL-C level(International Standard Unit: mmol/L) | 57 days
  Safety and tolerability will be assessed by the incidence and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
To assess the pharmacokinetic characteristics and dose proportionality relathionship of HST101 following a single SC dose | 57 days
  The PK parameters include Cmax, Tmax, T1/2, AUC0-t, AUCinf and others if necessary
To assess the PD effect of a single SC dose of HST101 on serum unbound (free) PCSK9 concentrations and serum LDL-C concentrations | 57 days
  Serum free PCSK9 and LDL-C will be measured at baseline and various time points over 57 days
To assess the effect of a single SC dose of HST101 on blood lipids including TC, HDL-C, VLDL-C, and TG | 57 days
  Serum TC,HDL-C,VLDL-C and TG（ISU:mmol/L）will be measured at baseline and various time points over 57 days to assess percent change from baseline over time
To assess the effect of a single SC dose of HST101 on serum ApoB, Apo A1 concentrations | 57 days
  Serum Apo B(ISU:mg/dL) , Apo A1(ISU:mg/dL) concentrations will be measured at baseline and various time points over 57 days to assess percent change from baseline over time
To assess the effect of a single SC dose of HST101 on serum Lp(a) concentrations | 57 days
  Serum Lp (a)(ISU: nmol/L) concentrations will be measured at baseline and various time points over 57 days to assess percent change from baseline over time
To assess the PK-PD relationship following a single SC dose of HST101 | 57 days
  The PK-PD relationship will be measured over 57 days
To assess immunogenicity (incidence, titer, and duration of ADAs/NAbs) following a single SC dose of HST101 | 57 days
  Measurement of ADAs/NAbs will be done at baseline and various intervals after HST101 administration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No